CLINICAL TRIAL: NCT04061460
Title: Respective Effects of Periodontal Oral Hygiene Instructions and Non-surgical Treatment on Clinical and Patient Related Outcomes: a Controlled Study in Non Smoker, Former Smoker and Smoker
Brief Title: Periodontal Treatment in Non Smokers, Former Smokers and Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Leila Salhi, principal investigator, head of clinic,Department of Periodontology, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B707201421977
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Periodontitis
Keywords: smoking; oral hygiene
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Intervention Model Description: at baseline, patients recieved oral hygiene instructions The same examiner (LS) performed an oral demonstration including teeth brushing, interdental cleaning and tong wash. Each patient received proper head and interdental brushes demonstration, moreover, patients were educated to brush their ventral face of their tong A single periodontist (L.S) performed the supra gingival debridment at the second appointment (2 weeks after receiving OHI) , followed 2 weeks after by a full month debridement using ultrason piezoelectric device (Newtron P5 XS Bled, Acteon, Satelec , France) with specific micro-inserts (H1, H3, H4L, H4R)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non smokers (Other): patient who never smoked
  Interventions: Procedure: mechanical plaque control
- former smoker (Other): patient who smoked in the past
  Interventions: Procedure: mechanical plaque control
- smoker (Other): patient who still smoke
  Interventions: Procedure: mechanical plaque control

INTERVENTIONS:
Procedure: mechanical plaque control — supra and sub gingival debridment ( plaque control)

SUMMARY:
The present study was designed as a prospective controlled study focusing on the effect of oral hygiene instructions and periodontal nonsurgical treatment( PNST) on clinical outcomes and patients related outcomes (PROMs) in smokers versus former smokers versus non smoker patients.

DETAILED DESCRIPTION:
75 consecutive patients presenting chronic periodontitis and who needed periodontal treatment were recruited in the Department of Periodontology and Oral Surgery at the University Hospital of Liège, Belgium (CHU, Sart-Tilman) according to the inclusion criteria.

The patients were subdivided between three groups: non-smoker (25), former smoker (25), and smoker patients(25).

Patients received informations about periodontitis genesis, the demonstration of oral hygiene instructions (OHI), the goal of PNST and the follow-up time were given ( baseline, after OHI, 3 months after PNST).

Periodontal clinical parameters and PROMS were collecetd and compared between 3 groups, at each visit.

Data collection:Periodontal clinical measurements and PROMS

The periodontal examination was conducted by a single periodontist (L.S) and included: probing depth (PD), gingival recession (RD), clinical attachment level (CAL), bleeding on probing (BOP), plaque score index (PI), Furcation (Furc), tooth mobility , the percentage of sites of PD ≥ 6mm and the number of missing tooth was recorded A graduated manual periodontal probe was used to take measurements at the 6 sites of each tooth. BOP (%) and plaque score (%) were collected as well as tooth mobility with a score from 1 to 3 . The furcation impairments were diagnosed with a Nabers probe according to the classification of Hamp and the Inflamed Surface Area (PISA) was calculated. Patients were classified according to the new periodontal classification identifying the grade, the stage and the extend of the periodontitis.

Patient-reported outcome measures (PROMs) A questionnaire using a visual analogue scale (VAS) was given to all participants regarding their oral hygiene habits, and perception about oral esthetic. The following questions were subjected to the patients: nine questions graduated scale from 0 to 10: 1/"How do you judge your degree of oral hygiene?", 2/"What is the frequency of utilization of interdental brushing?", 3/"Do you like the color of your teeth? , 4/"Your teeth are there sensitive to cold? , 5/ "How do you judge your degree of gingival health? , 6/ "How do you judge the esthetic aspect of you gum?", 7/ "Do you like the color of your gum? ", 8/ "Does your gum bleed during brushing?", 9/ "How do you judge your breath?".

sample size: The study was powered to detect a minimum clinically significant difference in probing depth (PD) of 0.5 mm between patients, using α= 0.05. The probing depth at baseline was considered covariate.

ELIGIBILITY:
Inclusion Criteria:

* aged of minimum 18 years old
* chronic periodontitis
* presence of a minimum of 6 teeth at each arch
* a minimum of 6 teeth with pocket depth of 5 mm
* signed the informed consent

Exclusion Criteria:

* aggressive periodontitis
* diabetes
* connective tissue disease
* pregnancy
* radio-therapy
* chemotherapy
* psychological disease
* previous periodontal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of probing depth (PD) | 2 weeks after baseline and 3 month after PNST
  PD was measured , in millimetern with periodontal probe, at 6 sites of each tooth

SECONDARY OUTCOMES:
Change from baseline of BOP (bleeding on probing) | 2 weeks after baseline and 3 month after PNST
  BOP was measured , in percentage of bleeding, at 6 sites of each tooth

IPD SHARING:
Plan to Share IPD: Undecided